CLINICAL TRIAL: NCT06973993
Title: The MORAL (MOzart Recorded And Live) Impact of Classical Music on Perceived Waiting Time and Satisfaction: A Comparative Study in Emergency Department Patients
Brief Title: A Study to Evaluate the Impact of Classical Music on Perceived Waiting Time and Satisfaction in Emergency Department Patients
Acronym: MORAL
Status: Recruiting | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Other Study IDs: ORBV-CHIR-006
Record Dates: First submitted 2025-04-11; First posted 2025-05-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Emergency Room
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- live music: All patients and relatives arriving at the ER on a given day will find live music as situation chosen in advance
  Interventions: Other: live music
- recorded music: All patients and relatives arriving at the ER on a given day will find recorded music as situation chosen in advance
  Interventions: Other: recorded music
- no music: All patients and relatives arriving at the ER on a given day will find no music as situation chosen in advance
  Interventions: Other: no music

INTERVENTIONS:
Other: live music — live music will be played during waiting time in ER room
  Groups: live music
Other: recorded music — recorded music will be transmitted during waiting time in ER room
  Groups: recorded music
Other: no music — no music will be played or transmitted during waiting time in ER room
  Groups: no music

SUMMARY:
The goal of this study is to evaluate whether classical music in the Emergency waiting room can diminish perception of waiting times. Patients and relatives, after arriving in the ER waiting room will either listen to live classical music, recorded classical music, or no music at all.

DETAILED DESCRIPTION:
The study was submitted to the ethics committee as an interventional clinical trial; however, they advised that it does not qualify as a clinical trial. The project does not collect health-related information from patients, according to the definition provided by swiss research law, and therefore does not require any authorization. They qualify it as a quality control initiative.

Please advise on how we should register it into clinicaltrials.gov, we might need the ID for publication purpose.

Thank you

ELIGIBILITY:
Inclusion Criteria:

* ER department patients waiting for medical assessment and their relatives
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Patients in situations of high severity and that pose an immediate significant threat to life or physiologic function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient and relatives affering ER
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | day 1
  Patient satisfaction will be calculated attributing a score to a validated questionnaire designed for assessing waiting times in the emergency department, namely the "Patient Satisfaction with Waiting Time in Emergency Departments" questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale Bellinzona e Valli, Ente Ospedaliero Cantonale, Bellinzona, Switzerland